CLINICAL TRIAL: NCT06312358
Title: Centering Community Partnerships to Facilitate Scaling Up of Infant Achievements for Community Implementation
Brief Title: Expanding the Infant Achievements Intervention Through Community Partnerships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rebecca Landa, Vice President, Professor, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00408654
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Child Development; Infant Development; Developmental Delay; Language Development
Keywords: Teacher Training; Mentoring; Inservice Training
MeSH Terms: conditions — Learning Disabilities | interventions — Capacity Building; Child Care

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to the study intervention consisting of (1) a professional development workshop and (2) weekly job-embedded coaching sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Teacher Professional Development Workshop and Coaching (Experimental): Teachers will participate in a professional development workshop session (approximately 2 hours in duration) followed by 8 weekly coaching sessions (approximately 45-60 minutes in duration). The study team (trained coaches) will utilize the Practice-Based Coaching model (Snyder et al., 2015) to support teachers' use of developmentally appropriate practices in early childhood classrooms. Teachers will be coached to implement strategies that foster responsive and nurturing relationships with young children.
  Interventions: Behavioral: Building Capacity for Infant Achievements in Child Care

INTERVENTIONS:
Behavioral: Building Capacity for Infant Achievements in Child Care — All teacher participants will be assigned to the professional development intervention consisting of an interactive workshop and weekly coaching sessions.

SUMMARY:
The goal of the research study is to increase teachers' implementation of evidence-based practices in Early Head Start classrooms through the delivery of a professional development (PD) training intervention. The main questions that the study aims to answer are:

1. Does teacher participation in a PD intervention improve the use of evidence-based practices from pre- to posttest?
2. To what extent is the PD intervention feasible to implement in an established child care program?
3. To what extent is the PD program acceptable to teachers?

Participants will attend PD workshops and participate in content-related job-embedded coaching sessions during the implementation of the study.

DETAILED DESCRIPTION:
The primary objective of the research study is to increase teachers' implementation of evidence-based practices in Early Head Start classrooms through the delivery of a professional development (PD) training intervention. It is hypothesized that teachers' fidelity to developmentally-appropriate practices, assessed through classroom observation measures, will increase following their participation in a comprehensive PD training intervention. The secondary hypotheses are that (1) the PD intervention is feasible to implement in an established child care program, and (2) the PD program is acceptable to teachers. Teacher participants will attend PD workshops, co-developed with community partners, and engage in follow-up job-embedded coaching sessions occurring weekly in their classrooms.

ELIGIBILITY:
Inclusion Criteria:

* Participants must currently work in an early childhood classroom serving children between 8-36 months of age.
* Participants must work in the role of a teacher or teacher assistant in an Early Head Start location.
* Participants must be willing to participate in two 60-90-minute trainings/workshops.
* Participants must be willing to participate in eight follow-up job-embedded coaching sessions

Exclusion Criteria:

* Works in a childcare setting outside of the Baltimore metro area
* Non-English speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Classroom Quality (as assessed by scores on the TPITOS) | Change from baseline/pretest up to posttest, up to 16 weeks.
  Classroom quality will be measured by total scores (ranging from 0-100%) on the Teaching Pyramid Model Infant-Toddler Observation Scale (TPITOS) which assesses the extent to which an early childhood program's staff is fostering responsive, nurturing relationships with young children and promoting strong social-emotional development.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, Principal Investigator — Kennedy Krieger Institute, Johns Hopkins University
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No